CLINICAL TRIAL: NCT00779012
Title: Post-Registration Open-Label, Non-Comparative, Multicenter Study of Rate of Efficacy and Tolerance of the Use of Anti-TNF Chimeric Monoclonal Antibodies (Remicade) in Treatment of Patients With Active Ankylosing Spondylitis
Brief Title: A Study of the Efficacy and Tolerance of Remicade in the Treatment of Active Ankylosing Spondylitis (Study P04042)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04042
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remicade (Experimental)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Remicade 5 mg/kg, given as an intravenous infusion over a 2-hour period followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 6 to 8 weeks (maximum 9 infusions).
  Other Names: Remicade; SCH 215596

SUMMARY:
The objective of this study is to prove reasonability of registration in Russian federation this new indication (ankylosing spondylitis [AS]) through evaluation of safety and efficacy rate of Remicade 5mg/kg, given as an intravenous infusion over a 2-hour period followed by additional 5 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 6 to 8 weeks (maximum 9 infusions).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 70 years of age.
* Males and female patients of reproductive potential (also includes women who have been postmenopaused <1 year) must use a reliable birth control method (abstinence, oral contraceptives, diaphragm prescribed by a physician, condom used with a spermicide, surgical sterilization) up until 6 months after the last Remicade infusion.
* Proven AS according to the modified New York criteria implying that included patients must have a pelvic x-ray showing the signs of sacroiliitis > grade 2 bilateral.
* Acute phase of disease during not less than last 3 months under condition of the everyday intake of some of NSAIDs in full daily dosage for at least 1 month before the initiation of the treatment, significant spinal pain (VAS > 4)during the last week prior to the inclusion into the study. In case of peripheral joints arthritis besides the measures mentioned above the absence of the efficacy of at least 2-times intraarticular injection of steroids (if only it is not contraindicated or not well tolerated) or sulfasalazine intake at a daily dose of 2-3 g for at least 4 months (if only it is not contraindicated or not well tolerated) should be established. In case of enthesitis inflammation besides the measures mentioned above the absence of the efficacy of at least 2-times local injection of steroids (if only it is not contraindicated or not well tolerated) should be established.
* Ability to comprehend the terms of the participation in the study, willing to follow all procedures and instructions and informed consent form signed before the beginning of the first procedures of the study (except several cases of chest x-ray).
* Screening for prevention of latent and active TB must be performed according to the local guidelines and/or the current SPC and alert card. This will include a PPD test and a Chest x-ray to be performed within 30 days prior to initiating treatment with Remicade.

Exclusion Criteria:

* Pregnant women, nursing mothers or a planned pregnancy within 6 months after the last infusion.
* Patients who have any concurrent systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from Remicade, e.g. Lyme disease, or a rheumatic disease (lupus erythematosus, systemic scleroderma) with the joint affection and sacroileitis.
* Prior administration of Remicade or any other therapeutic agent targeted at reducing TNF (e.g.,Etanercept, pentoxifylline, thalidomide or anti-CD4+ antibody) within the previous 3 months.
* History of known allergies to murine proteins.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute upper respiratory tract infection (colds) or uncomplicated urinary tract infection need not be considered exclusions at the discretion of the treating physician.
* Any chronic infections in the acute phase, e.g. upper respiratory tract infections or other localization (chronic bronchitis, pneumonia, pyelonephritis, cholecystitis, hepatitis etc.).
* Documented HIV infection.
* Positive hepatitis B and C test without clinical signs of the disease.
* Current skin psoriasis, nonspecific ulcerative colitis and Crohn's disease.
* History of opportunistic infections such as herpes zoster within 2 months of screening. Evidence of active CMV, active pneumocystis carinii, drug resistant atypical mycobacterium infections, etc.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past 5 years.
* Active and/or latent TB or previous history of TB.
* Non-stable doses of the basic steroid therapy or NSAID therapy within 4 weeks before the inclusion into the study.
* Supportive prednisone therapy >10 mg/day.
* Patients with moderate or severe heart failure (NYHA class III/IV).
* Septic arthritis (or infected joint implant) within at least last 12 months.
* Necessity in the use of other medicinal products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy and safety rate of the study drug, Remicade, in decreasing symptoms and signs of AS (pain) as well as the evaluation of the safety and the tolerance of the profile of the drug. | The patient undergoes the complex evaluation of the articular status every 6 -8 weeks.

SECONDARY OUTCOMES:
Frequency of achievement of at least 50% ASAS improvement (compared to baseline) 8 weeks after the last infusion of Remicade. | 8 weeks after the last infusion of Remicade
Frequency of at least 50% of the stable improvement of ASAS (compared to baseline) over a period of the supportive treatment phase (after infusion 3, up to 6 to 8 weeks after the last infusion of Remicade) | Up to 8 weeks after the last infusion of Remicade
Frequency of at least 20%, 50%, and 75% of ASAS improvement (compared to baseline) 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change in AS activity (BASDAI) compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of global evaluation of the activity of the disease by patient (VAS) compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of the functional status of the patients (BASFI) compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of spine motion compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of spinal pain compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of sensation of fatigue compared to baseline 6 to 8 weeks after the last infusion of Remicade (VAS) | Up to 8 weeks after the last infusion of Remicade
Change of pain in peripheral joints compared to baseline 6 to 8 weeks after the last infusion of Remicade (VAS) | Up to 8 weeks after the last infusion of Remicade
Change of the duration of the morning stiffness in peripheral joints compared to baseline 6 to 8 weeks after the last infusion of Remicade (VAS) | Up to 8 weeks after the last infusion of Remicade
Change of the number of tender joints compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of the number of inflamed joints compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of the number of the transformed enthesitises compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of the duration of the morning spinal stiffness compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Change of serum C-reactive protein and ESR compared to baseline 6 to 8 weeks after the last infusion of Remicade | Up to 8 weeks after the last infusion of Remicade
Quality of life evaluation in accordance with SF-36 | 6-8 weeks after visit 10 (before the last infusion of Remicade) or in case of discontinuation
Obtaining of additional information on the safety profile of the tested product over a period of the study. | up to 54 weeks

REFERENCES:
- [Result] Bunchuk NV, Rumiantseva OA, Loginova EIu, Bochkova AG, Storozhakov GI, Ettinger OA, Kosiura SD, Kamalova RG, Valishina LM. [The efficacy and safety of infliximab in patients with ankylosing spondylitis: results of an open-labeled multicenter study]. Ter Arkh. 2010;82(10):41-6. Russian. PMID 21341463
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html